CLINICAL TRIAL: NCT06850272
Title: Brisk Walking Training Compared with Cognitive Behavioral Therapy for the Treatment of Chronic Primary Insomnia in People Aged 60 Years or Above: a Randomized, Partially Blinded, Non-inferiority Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Zixin Wang, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECS24610123
Record Dates: First submitted 2025-02-23; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Primary Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brisk walking group (Experimental): Participants in the brisk walking training group receive an eight-week instructor-led interval brisk walking training (40 minutes/session, three sessions/week).
  Interventions: Behavioral: Brisk walking
- CBT-I group (Active Comparator): Participants in the CBT-I group receive standard-of-care group-based eight-session CBT-I (one session/week).
  Interventions: Behavioral: Cognitive-behavioral therapy for insomnia

INTERVENTIONS:
Behavioral: Brisk walking — Participants in the brisk walking training group receive an eight-week instructor-led interval brisk walking training (40 minutes/session, three sessions/week).
  Arms: Brisk walking group
Behavioral: Cognitive-behavioral therapy for insomnia — Participants in the CBT-I group receive standard-of-care group-based eight-session CBT-I (one session/week).
  Arms: CBT-I group

SUMMARY:
This study is a single-blinded (outcome assessor) and parallel-group non-inferiority RCT. Chinese older adults aged ≥60 years with chronic primary insomnia will be randomized evenly (1:1) to either the brisk walking training group or the CBT-I group. Participants in the brisk walking training group receive an eight-week instructor-led interval brisk walking training (40 minutes/session, three sessions/week). Participants in the CBT-I group receive standard-of-care group-based eight-session CBT-I (one session/week). Self-reported and objective sleep outcomes are measured at baseline (T0), after completion of the intervention (T1), and six (T2), and 12 months after T1 (T3).

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥60 years;
2. Ethnic Chinese; able to read, write and speak Cantonese
3. Having a Hong Kong ID;
4. Willing to wear an accelerometer on the wrist for a week to assess sleep parameters at T0, T1, and T2.
5. Score ≥10 in the Insomnia Severity Index (ISI) (presence of insomnia)
6. Experiencing any one of the following symptoms for ≥3 days per week

   1. Difficulty initiating sleep; OR
   2. Difficulty maintaining sleep; OR
   3. Early-morning awakening with inability to return to sleep

Exclusion Criteria:

1. Score ≥1 in the Chinese version of the Physical Activity Readiness Questionnaire (PAR-Q);
2. Currently regularly practicing a moderate-intensity PA program such as brisk walking or Tai Chi (≥3 times a week, ≥30 minutes/session);
3. Currently receiving or scheduled to receive CBT-I during the study period;
4. Score ≤16 in the validated telephone version of the Cantonese Mini-Mental State Examination (T-CMMSE).
5. Working nightshifts and unable/unwilling to discontinue such work pattern;
6. Having a diagnosis of a major depressive disorder, anxiety disorders or other severe mental disorder (bipolar disorders, psychosis). Those with mild depression or anxiety disorders will not be excluded;
7. Use of antidepressant or antipsychotic medication or under treatment of other serious diseases (e.g., cancer chemotherapy) known to affect sleep;
8. Presence of any serious chronic diseases which affect sleep (e.g., cancer, autoimmune diseases).
9. Having a serious somatic condition preventing the participation of brisk walking training/CBT-I.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Score of the Insomnia Severity Index (ISI) | 12 months
  Score of the Insomnia Severity Index (ISI) measured at at baseline (T0), after completion of the intervention (T1), and six (T2), and 12 months after T1 (T3).

SECONDARY OUTCOMES:
Insomnia remission | 12 months
  Structured clinical interview to confirm insomnia remission based on the DSM-5 criteria at 12 months after completion of the intervention
Sleep quality | 12 months
  Sleep quality will be measured by the 19-item Pittsburg Sleep Quality Index (PSQI) at baseline (T0), after completion of the intervention (T1), and six (T2), and 12 months after T1 (T3)
Seven-day ActiGraph | 12 months
  Seven-day ActiGraph at baseline (T0), after completion of the intervention (T1), and six (T2), and 12 months after T1 (T3)

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The individual participant data contains sensitive behaviors and conditions.